CLINICAL TRIAL: NCT00342251
Title: Age-Related Macular Degeneration: A Genetic Epidemiology Study in the Amish
Brief Title: Investigating Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903235; 03-EI-N235
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-04

CONDITIONS: Age-Related Macular Degeneration
Keywords: Macular Degeneration; Retinal Images; Risk Factors; Linkage Analysis; Gene; Mutation
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Age-related macular degeneration (ARMD) affects older Americans and can lead to irreversible blindness. Although the cause if ARMD is unclear, it appears to be a condition that is affected by both genetic and environmental influences.

The purpose of this study is to examine an Amish community to investigate genetic factors in the development of ARMD.

Study participants will be 1,000 members, ages 50 and older, of the Old Order Amish community in Lancaster and Franklin counties in Pennsylvania. Each will undergo a 30-minute dilated eye exam during which an ophthalmologist or optometrist will take digital images of the macula and optic disc. Depending on the results of their eye exam, participants may be asked to give a blood sample as well. They will also complete a brief questionnaire about personal exposure related to occupation, sunlight and smoking.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a leading cause of visual impairment in the United States. Available evidence suggests that AMD is a complex disorder with a significant genetic component as well as potential environmental influences. In this study we propose to examine 3,000 members, ages 50 and older, of the Old Order Amish community in the Lancaster and Franklin counties area in Pennsylvania. We plan to detail the epidemiology of AMD in this population isolate in attempt to elucidate genetic factors which may confer susceptibility and predispose some Amish individuals and their families to develop AMD. All study participants agreeing to enroll and providing informed consent will undergo a complete, dilated eye examination during which digital stereo images of the macula and optic disc regions will be acquired. Study participants will also be asked to complete a brief questionnaire inquiring about personal exposures related to occupation, sunlight, and smoking. AMD will be determined by an independent reading of the digital fundus photographs by the University of Wisconsin Fundus Photography Reading Center according to the AREDS AMD classification scheme. We will employ standard statistical genetics methods of parametric and non-parametric linkage analysis, association analysis, and transmission disequilibrium tests, with allowances for environmental (i.e. non-genetic) factors to determine if we can identify any candidate regions or candidate genes that predispose Amish individuals to an increased risk of AMD. Ultimately, we hope to follow up any regions that show suggestive evidence of linkage on the genome-wide scan with fine mapping in those regions, leading to eventual cloning and sequencing of a gene or genes.

ELIGIBILITY:
* INCLUSION CRITERIA:

All Amish individuals, ages 50 and older, who either respond in the affirmative to the letter of invitation or are self-referred to the Amish clinic for participation in the AMD study, will be eligible.

EXCLUSION CRITERIA:

Individuals who decline participation, who are unwilling to sign the Consent Form, and who are not recognized by the Amish as being Amish will be excluded.

There are no clinical inclusion/exclusion criteria.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2003-06-20; Study Completion 2012-04-04

CONTACTS AND LOCATIONS:
Overall Officials: Susan Vitale, Ph.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States